CLINICAL TRIAL: NCT00117273
Title: A Prospective, Single-Center, Open-Label, Randomized Study to Evaluate Suppression of the Pituitary-Ovarian Axis With Three Different Regimens of Oral Contraceptive Pills
Brief Title: A Study to Evaluate Suppression of the Pituitary-Ovarian Axis With Three Different Oral Contraceptive Regimens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR PSE 310
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — Seasonale; Levonorgestrel; Seasonique; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Seasonique (LNG/EE and EE)
- 2 (Active Comparator)
  Interventions: Drug: Seasonale [levonorgestrel (LNG)/ethinyl estradiol (EE)]
- 3 (Active Comparator)
  Interventions: Drug: Portia (LNG/EE)

INTERVENTIONS:
Drug: Seasonale [levonorgestrel (LNG)/ethinyl estradiol (EE)] — 1 tablet daily
  Arms: 2
Drug: Seasonique (LNG/EE and EE) — 1 tablet daily
  Arms: 1
Drug: Portia (LNG/EE) — 1 tablet daily x 28 days
  Arms: 3

SUMMARY:
This is a randomized, open-label study to evaluate pituitary ovarian suppression in healthy, reproductive-aged women using three different regimens of oral contraceptives (OCs). Two extended regimen OCs, Seasonale (levonorgestrel/ethinyl estradiol 0.15/0.03 mg for 84 days followed by 7 days of placebo), and Seasonique (levonorgestrel/ethinyl estradiol 0.15/0.03 mg for 84 days followed by 7 days of ethinyl estradiol 0.01 mg), and a 28-day regimen OC, Portia (levonorgestrel/ethinyl estradiol 0.15/0.03 mg for 21 days followed by 7 days of placebo).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Not pregnant or breastfeeding
* Weight <200 lbs
* Currently taking oral contraceptives in the standard 28-day regimen for at least two months

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Pregnancy within the last 3 months
* Smoking > 10 cigarettes per day

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Compare differences in hormone patterns (follicle stimulating hormone [FSH], luteinizing hormone [LH], inhibin-B, and estradiol) | Before, during and after the 7-day hormone free interval or EE-supplemented interval

SECONDARY OUTCOMES:
Compare the differences in hormone withdrawal symptoms | Before, during and after the 7-day hormone free interval or EE-supplemented interval
Compare differences in ovarian follicular development | Before, during and after the 7-day hormone free interval or EE-supplemented intervals

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (1):
- Duramed Investigational Site, Temple, Texas, United States

REFERENCES:
- See also: Mayo Clinic - Birth Control Guide — http://www.mayoclinic.com/health/birth-control/BI99999